CLINICAL TRIAL: NCT07140770
Title: Sleep and Physical Activity in Patient and Caregiver Dyads Following Allogeneic Hematopoietic Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0317; NCI-2025-06207 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Physical Activity; Sleep; Allogenic Hematopoietic Cell Transplant
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fitbit — You will wear the tracker on your wrist like a watch and it will continuously (non-stop) monitor your activity, sleep, and heart rate.
  Functional testing will be completed with a research team member and will consist of 2 tests: testing your grip strength by having you squeeze a measuring device 3 times with your dominant hand and measuring how many minutes it takes for you to walk 15 feet.
Other: Questionnaire — Complete questionnaires at 3 timepoints, at the time of enrollment on the day of allogeneic hematopoietic cell transplantation, 8 days after allogeneic hematopoietic cell transplantation, and 7 days after hospital discharge.

SUMMARY:
To understand the changes in health-related quality of life of patients and caregivers after allogeneic hematopoietic cell transplantation.

DETAILED DESCRIPTION:
Primary Objectives

* Assess the feasibility and acceptability of obtaining objective sleep and physical activity measures in participants receiving allogeneic HCT and their caregivers during hospitalization (T2), and after discharge (T3) using Fitbits.
* Feasibility will be determined by the percentage of participants and caregivers who wear the Fitbit Inspire 3 for sleep and physical activity data at T2, and T3. For the purposes of this study, if ≥70% of participants and caregivers will wear the Fitbit for 5 of 7 nights for sleep data and at least 10 hours during waking hours for 5 of 7 days for physical activity data at both data collection periods, the study will be determined to be feasible. Feasibility will be reported for participants and caregivers separately and will include the percentage of eligible participants who are approached, agree to participate, and complete research activities.

Secondary Objectives

* Examine trends in objectively measured sleep, physical activity, and frailty, and participant-reported sleep disturbance, sleep-related impairment, anxiety, depression, fatigue, cancer treatment distress, and quality of life in allogeneic HCT participants and their caregivers during hospitalization (T2), and after discharge (T3).
* Hypothesis 1: HCT participants will demonstrate improvements in objectively measured sleep, physical activity, and frailty, and participant-reported sleep disturbance, sleep-related impairment, anxiety, depression, fatigue, and cancer treatment distress from T2 to T3.
* Compare objectively measured sleep and physical activity, and participant-reported sleep disturbance, sleep-related impairment, anxiety, depression, fatigue, cancer treatment distress, and quality of life between allogeneic HCT participants and their caregivers during hospitalization (T2), and after discharge (T3).
* Hypothesis: HCT participants will demonstrate significant improvements compared to their caregivers in objectively measured sleep and physical activity, and patient-reported sleep disturbance, sleep-related impairment, anxiety, depression, fatigue, cancer treatment distress, and quality of life.
* Acceptability will be assessed using an investigator-developed instrument, the Physical Activity and Sleep Tracker Acceptability Survey.

ELIGIBILITY:
Eligibility Criteria

* Participants and caregivers ages 18 years and older.
* Participants diagnosed with a hematologic malignancy with a scheduled allogeneic HCT.
* Caregivers identified by participant as the primary caregiver.
* Participants and caregivers able to read, speak, and consent in English.
* Participants and caregivers able to understand and be willing to sign a written informed consent document.
* Participants and caregivers must have internet access via smart phone or tablet with the capacity to 1) download the Fitbit app and 2) complete study assessments with study

Exclusion Criteria

* Participant or caregiver unable to provide consent, such as cognitively impaired individuals
* Participant or caregiver with a diagnosis of sleep apnea.
* Primary caregiver is a paid professional, such as a live-in Registered Nurse.
* Participant has multiple caregivers and is unable to identify one primary caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | Through study completion; an average of 1 year
  You will answer questionnaires with a member of the research team. The questionnaires will take about 35 minutes complete. You will be asked questions about your sleep, anxiety and depressive symptoms, fatigue, distress, and your quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen D Hacker, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org